CLINICAL TRIAL: NCT01709708
Title: Use of the Tx360 Nasal Applicator for Transnasal Sphenopalatine Ganglion Block in the Treatment of Chronic Migraine: A Double-blind Placebo-controlled Study
Brief Title: Use of the Tx360 Nasal Applicator in the Treatment of Chronic Migraine
Acronym: Tx360
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tian Medical Inc. (Industry)
Collaborators: Clinvest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-004TI
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Chronic Migraine
Keywords: Migraine; Headache; Chronic Migraine; Marcaine; Tx360
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Bupivacaine; Drugs, Generic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Marcaine (Active Comparator): Group A will receive treatment with 0.3 mL of 0.5% Marcaine delivered bilaterally with the Tx360™ device to the mucosa associated with the Sphenopalatine Ganglion (SPG)
  Interventions: Drug: Marcaine
- Saline (Placebo Comparator): Group B will receive saline placebo delivered bilaterally with the Tx360TM device to the mucosa associated with the SPG.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Marcaine — Marcaine used as a topical local anesthetic to block the SPG by delivering Marcaine directly to the specific area of mucosa associated with the SPG.
  Other Names: Bupivicane (generic)
  Arms: Marcaine
Drug: Saline — Saline
  Arms: Saline

SUMMARY:
Migraine imposes a substantial burden on patients in terms of diminished daily functioning, quality of life, and financial loss. Pain severity and duration correlates with reduced measures of daily functioning, and overall health status. The sphenopalatine ganglion (SPG) has been implicated in a variety of cephalalgias. This has been well represented in the literature dating back over a century. Access to this structure can be gained via a small area of mucosa just posterior and superior to the tail of the middle turbinate on the lateral nasal wall. At this aspect, there is no bony boundary to the SPG. Blocking the SPG using local anesthetics relieves pain. Unfortunately, many current interventions are cumbersome, invasive, and expensive. The purpose of this study is to evaluate the efficacy of the Tx360™, a new nasal applicator device, in the treatment of head and face pain and to examine the economic implications. The Tx360™ is a single use device designed to deliver a topical local anesthetic to the specific area of mucosa associated with the SPG. A total of 42 study participants will be accepted into this double-blind placebo-controlled study. 28 will receive SPG blocks using a 0.3 mL of a 0.5% solution of Marcaine delivered by the Tx360™ while 14 will receive a placebo of saline substituted for the Marcaine. Both patient sets will also be given a piece of lemon hard candy as a taste distractor. Participants must have a chronic migraine history with over 15 symptomatic days per month over the past three months. The treatment plan consists of six weeks of treatment, two times per week. Short and longer term assessments will be retrieved and analyzed as detailed in the Study Design.

DETAILED DESCRIPTION:
42 study participants will be included in this double-blind placebo-controlled study. Following enrollment of 42 subjects and completion of the 6-week Treatment Period by all active subjects, an analysis of the treatment effect will be performed for a reassessment of sample size and, if deemed appropriate, the study will continue with enrollment of additional subjects to ensure a more statistically robust interpretation of the data. The results of the statistical analysis will be blinded from Investigators and coordinators. The procedure will be delivered to all subjects who agree to participate, meet inclusion criteria, and sign informed consent.

At Visit 1 following Informed Consent, a physical exam and vital signs will be completed. A medical, headache, and medication history (to include age, sex, height and weight, and duration and location of headache pain, as well as history of ER visits) will be collected on all subjects. Eligible subjects will be provided with a Baseline Headache Diary and instructed to treat migraines for the following month in their usual manner with their usual treatment. The daily Diary will document headache, acute treatment and response, and migraine associated symptoms (nausea, vomiting, light sensitivity, or sound sensitivity) to establish a Baseline number of headache days and severity. Visit 2 will be scheduled for 1 month following Visit 1. Following Visit 1, Visits 2-13 (treatment visits) will be scheduled to occur twice weekly (during the regular Monday - Friday work week) at least 2 days apart. Treatments should not occur on consecutive days.

At Visit 2, the Baseline Headache Diary will be reviewed and those subjects continuing to meet eligibility will be dispensed a 6-week Treatment Period Diary and complete Before Procedure questions to include the Pain Intensity Numeric Rating Scale (NRS), the Modified Pain Characteristic Questionnaire, and a baseline Headache Impact Test-6 (HIT-6), have vital signs completed, and the medical, headache, and medication history updated. Subjects will be randomized 2:1 to Group A or Group B. Group A will receive treatment with 0.3 mL of 0.5% Marcaine delivered bilaterally with the Tx360™ device to the mucosa associated with the SPG. Group B will receive saline substituted for Marcaine delivered bilaterally with the Tx360TM device to the mucosa associated with the SPG.

To maintain the blinding of the treatment groups, neither the Investigator nor research personnel who are involved in evaluating the subject should prepare the study medication. An independent research staff person with no involvement in the study conduct will place study medication (either Marcaine for a subject randomized to Group A or Placebo/saline for a subject randomized to Group B) in a 1cc Luer Lok tip syringe and assemble the syringe and Tx360TM catheter as instructed in training. A label with the subject Drug Number will be placed on the device at that time. The research staff person administering the study medication will verify that the Drug Number assignment is correct.

Both Groups will be given a piece of lemon hard candy as a taste distractor.

At each treatment visit (Visits 2-13), in addition to Before Procedure questions, subjects will complete 15-minute and 30-minute After Procedure questionnaires to include the NRS and, at 30 minutes, the Patient's Global Impression of Change (PGIC). Subjects will take home a questionnaire to include the NRS, PGIC, satisfaction question, and the Modified Pain Characteristic Questionnaire to be completed at 24 hours following treatment and be instructed to return the 24-hour After Procedure questionnaire to the clinic at the next visit.

At Visits 2-15 vital signs will be completed, medications will be updated, and Non-Serious Adverse Events will be collected after the first treatment. Serious Adverse Events will be collected once the informed consent has been signed and throughout the study.

At Visits 5, 8, and 11, the Treatment Period Headache Diary will be collected, reviewed, and re-dispensed.

At Visit 13, the 1-Month Post-Treatment Period Diary will be dispensed.

The subject will return to the clinic at Visit 14 between 24 and 96 hours following the final treatment at Visit 13 to return the 24-hour After Procedure Questionnaire and complete the 1-Month Treatment Period HIT-6. The Treatment Period Diary will be collected.

At Visit 15, 1 month following the final treatment, each subject will return to the clinic and complete a 1-Month Follow Up HIT-6 and the 1-Month Follow Up Questionnaire. The 1-Month Post-Treatment Period Diary will be collected.

At 6 months following the final treatment, each subject will be phoned to complete the 6-Month Follow Up Questionnaire to include the NRS, PGIC, satisfaction question, the Modified Pain Characteristic Questionnaire, and a 6-Month Follow Up HIT-6.

Treatment Medication Subjects randomized to Group A will be administered 0.3 mL of 0.5% Marcaine delivered bilaterally with the Tx360™ device to the mucosa associated with the SPG. Twelve treatments will be administered over a period of 6 weeks.

Subjects randomized to Group B will be administered saline substituted for Marcaine delivered bilaterally with the Tx360TM device to the mucosa associated with the SPG for treatment of chronic migraine. Twelve treatments will be administered over a period of 6 weeks.

Rescue Medication Subjects will be allowed to rescue with medication mutually agreed upon by subject and Investigator at the time of screening.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, in otherwise good health, 18 to 80 years of age.
2. Has history of chronic migraine (with or without aura) according to the criteria proposed by the Headache Classification Committee of the International Headache Society for at least 3 months prior to enrollment.
3. Has onset of migraine before age 50.
4. Is able to differentiate migraine from any other headache they may experience (e.g., tension-type headache).
5. Is not currently taking a migraine preventive or has been taking preventive for at least 30 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period.
6. If female of childbearing potential, agrees to use, for the duration of the study, a medically acceptable form of contraception as determined by the Investigator.

   1. Complete abstinence from intercourse from 2 weeks prior to administration of study drug throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the study drug; or,
   2. Surgically sterile (hysterectomy or tubal ligation or otherwise incapable of pregnancy); or,
   3. Sterilization of male partner; or,
   4. Intrauterine device with published data showing lowest expected failure rate is less than 1% per year; or,
   5. Double barrier method (i.e., 2 physical barriers OR 1 physical barrier plus spermicide) for a least 1 month prior to Visit 1 and throughout study; or,
   6. Hormonal contraceptives for at least 3 months prior to Visit 1 and throughout study.
7. Has pain presentation in frontal, temporal, ophthalmic, maxillary, mandibular, facial, or intraoral location.

Exclusion Criteria:

1. Is male or female, in otherwise good health, 18 to 80 years of age.
2. Has history of chronic migraine (with or without aura) according to the criteria proposed by the Headache Classification Committee of the International Headache Society for at least 3 months prior to enrollment.
3. Has onset of migraine before age 50.
4. Is able to differentiate migraine from any other headache they may experience (e.g., tension-type headache).
5. Is not currently taking a migraine preventive or has been taking preventive for at least 30 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period.
6. If female of childbearing potential, agrees to use, for the duration of the study, a medically acceptable form of contraception as determined by the Investigator.

   1. Complete abstinence from intercourse from 2 weeks prior to administration of study drug throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the study drug; or,
   2. Surgically sterile (hysterectomy or tubal ligation or otherwise incapable of pregnancy); or,
   3. Sterilization of male partner; or,
   4. Intrauterine device with published data showing lowest expected failure rate is less than 1% per year; or,
   5. Double barrier method (i.e., 2 physical barriers OR 1 physical barrier plus spermicide) for a least 1 month prior to Visit 1 and throughout study; or,
   6. Hormonal contraceptives for at least 3 months prior to Visit 1 and throughout study.
7. Has pain presentation in frontal, temporal, ophthalmic, maxillary, mandibular, facial, or intraoral location.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tian Xia, MD, Principal Investigator — Tian Medical Inc.
Locations (2):
- United States (2):
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Clinvest/A Division of Banyan Group, Inc., Springfield, Missouri

REFERENCES:
- [Background] Tepper SJ. A pivotal moment in 50 years of headache history: the first American Migraine Study. Headache. 2008 May;48(5):730-1; discussion 732. doi: 10.1111/j.1526-4610.2008.01117_1.x. PMID 18471125
- [Background] Piagkou M, Demesticha T, Troupis T, Vlasis K, Skandalakis P, Makri A, Mazarakis A, Lappas D, Piagkos G, Johnson EO. The pterygopalatine ganglion and its role in various pain syndromes: from anatomy to clinical practice. Pain Pract. 2012 Jun;12(5):399-412. doi: 10.1111/j.1533-2500.2011.00507.x. Epub 2011 Sep 29. PMID 21956040
- [Background] Oluigbo CO, Makonnen G, Narouze S, Rezai AR. Sphenopalatine ganglion interventions: technical aspects and application. Prog Neurol Surg. 2011;24:171-179. doi: 10.1159/000323049. Epub 2011 Mar 21. PMID 21422787
- [Background] Windsor RE, Jahnke S. Sphenopalatine ganglion blockade: a review and proposed modification of the transnasal technique. Pain Physician. 2004 Apr;7(2):283-6. PMID 16868606
- [Background] Rosenberg M, Phero JC. Regional anesthesia and invasive techniques to manage head and neck pain. Otolaryngol Clin North Am. 2003 Dec;36(6):1201-19. doi: 10.1016/s0030-6665(03)00134-8. PMID 15025017
- [Background] Wood PB. Role of central dopamine in pain and analgesia. Expert Rev Neurother. 2008 May;8(5):781-97. doi: 10.1586/14737175.8.5.781. PMID 18457535
- [Background] Boivie J. Chapter 48 Central post-stroke pain. Handb Clin Neurol. 2006;81:715-30. doi: 10.1016/S0072-9752(06)80052-7. No abstract available. PMID 18808870
- [Background] Stankewitz A, Voit HL, Bingel U, Peschke C, May A. A new trigemino-nociceptive stimulation model for event-related fMRI. Cephalalgia. 2010 Apr;30(4):475-85. doi: 10.1111/j.1468-2982.2009.01968.x. Epub 2010 Feb 1. PMID 19673914
- [Background] Herrera Tolosana S, Fernandez Liesa R, Escolar Castellon Jde D, Perez Delgado L, Lisbona Alquezar MP, Tejero-Garces Galve G, Guallar Larpa M, Ortiz Garcia A. [Sphenopalatinum foramen: an anatomical study]. Acta Otorrinolaringol Esp. 2011 Jul-Aug;62(4):274-8. doi: 10.1016/j.otorri.2011.01.009. Epub 2011 Mar 22. Spanish. PMID 21429469
- [Background] Rusu MC. Microanatomy of the neural scaffold of the pterygopalatine fossa in humans: trigeminovascular projections and trigeminal-autonomic plexuses. Folia Morphol (Warsz). 2010 May;69(2):84-91. PMID 20512758
- [Background] Oomen KP, Ebbeling M, de Ru JA, Hordijk GJ, Bleys RL. A previously undescribed branch of the pterygopalatine ganglion. Am J Rhinol Allergy. 2011 Jan-Feb;25(1):50-3. doi: 10.2500/ajra.2011.25.3550. PMID 21711979
- [Background] Siessere S, Vitti M, Sousa LG, Semprini M, Iyomasa MM, Regalo SC. Anatomic variation of cranial parasympathetic ganglia. Braz Oral Res. 2008 Apr-Jun;22(2):101-5. doi: 10.1590/s1806-83242008000200002. PMID 18622477
- [Background] Gronseth G, Cruccu G, Alksne J, Argoff C, Brainin M, Burchiel K, Nurmikko T, Zakrzewska JM. Practice parameter: the diagnostic evaluation and treatment of trigeminal neuralgia (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology and the European Federation of Neurological Societies. Neurology. 2008 Oct 7;71(15):1183-90. doi: 10.1212/01.wnl.0000326598.83183.04. Epub 2008 Aug 20. PMID 18716236
- [Background] Yang lY, Oraee S. A novel approach to transnasal sphenopalatine ganglion injection. Pain Physician. 2006 Apr;9(2):131-4. PMID 16703973
- [Background] Kanai A, Suzuki A, Kobayashi M, Hoka S. Intranasal lidocaine 8% spray for second-division trigeminal neuralgia. Br J Anaesth. 2006 Oct;97(4):559-63. doi: 10.1093/bja/ael180. Epub 2006 Aug 1. PMID 16882684
- [Derived] Cady RK, Saper J, Dexter K, Cady RJ, Manley HR. Long-term efficacy of a double-blind, placebo-controlled, randomized study for repetitive sphenopalatine blockade with bupivacaine vs. saline with the Tx360 device for treatment of chronic migraine. Headache. 2015 Apr;55(4):529-42. doi: 10.1111/head.12546. Epub 2015 Mar 31. PMID 25828648
- [Derived] Cady R, Saper J, Dexter K, Manley HR. A double-blind, placebo-controlled study of repetitive transnasal sphenopalatine ganglion blockade with tx360((R)) as acute treatment for chronic migraine. Headache. 2015 Jan;55(1):101-16. doi: 10.1111/head.12458. Epub 2014 Oct 23. PMID 25338927
- See also: Instructions for use and device training — http://www.tianmedical.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Marcaine | Saline
Started | 27 | 14
Completed | 26 | 12
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marcaine | Saline | Total
Number analyzed (Participants) | 27 | 14 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.96 (11.63) | 41.97 (14.71) | 41.30 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 11 | 31
  Male | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 20 | 14 | 34
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS)
Description: Compare Numeric Rating Scale (NRS) scores Before Procedure,15-Minute Post Treatment, 30-Minutes Post Treatment, 24-Hour Post Treatment for all 12 treatments (Marcaine vs. Saline). NRS is a likert scale ranging from 0-10 with 0 being no pain and 10 being worst possible pain. For each individual time point, all 12 treatments were averaged for that time point and a single value was used for comparison between the two groups.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
units on a scale
  Before Procedure | 3.18 (2.79) | 3.78 (2.48)
  15 Minutes Post Treatment | 2.53 (2.61) | 3.51 (2.39)
  30 Minutes Post Treatment | 2.41 (2.61) | 3.45 (2.36)
  24 Hours Post Treatment | 2.85 (2.74) | 4.20 (2.62)

2. Secondary Outcome: Change in Numeric Rating Scale (NRS)
Description: Compare percentage change in Numeric Rating Scale (NRS) score from Before Procedure to 15-Minutes, Before Procedure to 30-Minutes, Before Procedure to 24-Hours After Procedure for all 12 treatments (Mean of all 12 treatments for each timepoint, comparing Group A to Group B). NRS is a likert scale ranging from 0-10 with 0 being no pain and 10 being worst possible pain.
Time Frame: 15 Minutes Post Treatment, 30 minutes Post Treatment and 24 hours Post Treatment, assessed up to 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
percentage of change
  15 Minutes Post Treatment | -23.3 (34.5) | -4.31 (27.3)
  30 Minutes Post Treatment | -27.7 (37.1) | -5.41 (29.2)
  24 Hours Post Treatment | -15.5 (69.9) | 13.5 (78.8)

3. Secondary Outcome: Patient's Global Impression of Change (PGIC)
Description: Compare 24-Hour After Procedure Patient's Global Impression of Change (PGIC) score for 12 treatments (Mean of all 12 treatments for each timepoint, comparing Group A to Group B). PGIC is a likert scale ranging from 1 to 7 with 1 being very much improved and 7 being very much worse.
Time Frame: 30 minutes Post Treatment and 24 hours Post Treatment, assessed up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
units on a scale
  30 Minutes Post Treatment | 3.00 (1.02) | 3.72 (0.53)
  24 Hours Post Treatment | 3.08 (1.26) | 3.88 (1.02)

4. Secondary Outcome: Modified Pain Characteristic Questionnaire
Description: Compare Modified Pain Characteristic Questionnaire scores Before Procedure vs. 24-Hour After Procedure, Before Procedure vs. 1-Month Follow Up, and Before Procedure vs. 6-Month Follow Up (Mean of all 12 treatments for each timepoint, comparing Group A to Group B). The modified pain characteristic questionnaire is a series of 11 questions on a likert scale ranging from 0 to 10 with 0 being no pain or does not interfere and 10 being worst pain or completely interferes. Percentage questions range from 0 to 100.
Time Frame: Before Treatment, 24 Hours After Treatment, 1 Month Post Treatment, and 6 Months Post Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
units on a scale
  Worst Pain Question: Before Treatment | 4.75 (3.11) | 6.15 (2.65)
  Worst Pain Question: 24 Hours After Treatment | 4.36 (3.01) | 6.16 (2.44)
  Worst Pain Question: 1 Month Post Treatment | 4.56 (3.23) | 5.64 (3.04)
  Worst Pain Question: 6 Months Post Treatment | 4.27 (3.10) | 5.88 (1.73)
  Least Pain Question: Before Treatment | 2.01 (2.55) | 2.50 (2.13)
  Least Pain Question: 24 Hours After Treatment | 1.77 (2.49) | 2.43 (1.93)
  Least Pain Question: 1 Month Post Treatment | 1.88 (2.62) | 2.64 (2.11)
  Least Pain Question: 6 Months Post Treatment | 1.68 (2.03) | 2.88 (2.47)
  Average Pain Question: Before Treatment | 3.39 (2.61) | 4.33 (2.29)
  Average Pain Question: 24 Hours After Treatment | 3.07 (2.57) | 4.27 (2.09)
  Average Pain Question: 1 Month Post Treatment | 3.36 (2.87) | 3.91 (2.30)
  Average Pain Question: 6 Months Post Treatment | 2.86 (2.62) | 4.00 (2.27)
  Percent Relief Question: Before Treatment | 41.3 (36.5) | 29.2 (33.0)
  Percent Relief Question: 24 Hours After Treatment | 46.0 (38.2) | 29.8 (32.5)
  Percent Relief Question: 1 Month Post Treatment | 46.3 (39.9) | 21.0 (32.1)
  Percent Relief Question: 6 Months Post Treatment | 34.7 (29.2) | 18.6 (30.8)
  General Activity Question: Before Treatment | 2.49 (2.96) | 3.50 (2.70)
  General Activity Question: 24 Hours After Treatmen | 2.31 (2.90) | 3.64 (2.78)
  General Activity Question: 1 Month Post Treatment | 2.64 (2.91) | 3.91 (2.81)
  General Activity Question: 6 Months Post Treatment | 2.68 (2.87) | 4.00 (3.32)
  Mood Interference Question: Before Treatment | 2.57 (3.07) | 3.78 (2.84)
  Mood Interference Question: 24 Hours After Treatme | 2.42 (3.06) | 4.19 (3.04)
  Mood Interference Question: 1 Month Post Treatment | 2.96 (3.43) | 3.82 (3.40)
  Mood Interference Question: 6 Months Post Treatmen | 3.18 (3.26) | 5.71 (3.68)
  Walking Ability Question: Before Treatment | 0.63 (1.27) | 1.27 (2.24)
  Walking Ability Question: 24 Hours After Treatment | 0.54 (1.33) | 1.24 (2.37)
  Walking Ability Question: 1 Month Post Treatment | 0.80 (1.68) | 0.55 (0.93)
  Walking Ability Question: 6 Months Post Treatment | 0.45 (1.74) | 0.43 (1.13)
  Normal Work Question: Before Treatment | 2.53 (3.08) | 3.49 (2.81)
  Normal Work Question: 24 Hours After Treatment | 2.21 (3.02) | 3.63 (2.97)
  Normal Work Question: 1 Month Post Treatment | 2.52 (3.14) | 3.45 (2.94)
  Normal Work Question: 6 Months Post Treatment | 2.59 (2.77) | 3.71 (3.50)
  Relationships Question: Before Treatment | 2.00 (2.87) | 3.47 (2.92)
  Relationships Question: 24 Hours After Treatment | 1.96 (2.87) | 3.90 (3.09)
  Relationships Question: 1 Month Post Treatment | 2.36 (3.29) | 3.09 (3.45)
  Relationships Question: 6 Months Post Treatment | 2.05 (2.87) | 3.86 (3.98)
  Sleep Interference Question: Before Treatment | 2.29 (3.09) | 2.68 (3.11)
  Sleep Interfere Question: 24 Hours After Treatment | 1.89 (3.03) | 2.85 (3.22)
  Sleep Interferenc Question: 1 Month Post Treatment | 1.92 (3.00) | 2.55 (3.47)
  Sleep Interference Question: 6 Months Post Treatme | 1.55 (2.32) | 3.14 (3.93)
  Enjoyment Question: Before Treatment | 2.81 (3.24) | 3.12 (2.74)
  Enjoyment Question: 24 Hours After Treatment | 2.58 (3.29) | 3.34 (2.89)
  Enjoyment Question: 1 Month Post Treatment | 2.64 (3.51) | 3.09 (2.91)
  Enjoyment Question: 6 Months Post Treatment | 3.18 (3.36) | 4.00 (4.12)

5. Secondary Outcome: Migraine Headache Days
Description: Compare change in the number of migraine headache days per month reported in Baseline Period Diary vs. Treatment Period Diary vs. Post-Treatment Period Diary.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: Migraine headache days per month
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
Migraine headache days per month
  Baseline | 15.0 (6.33) | 15.8 (7.40)
  Treatment | 12.3 (8.83) | 12.2 (9.69)
  Post Treatment | 10.8 (9.22) | 11.3 (8.32)

6. Secondary Outcome: Acute Medications Usage
Description: Number of acute medications used during Treatment period (6 weeks) and Follow-Up (4 weeks) (Group A vs. Group B).
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: Number of medications used
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
Number of medications used | 29.3 (28.2) | 47.4 (54.2)

7. Secondary Outcome: Adverse Events
Description: Number of adverse events over the entire length of study (Group A vs. Group B).
Time Frame: 34 weeks
Measure: Mean (Standard Deviation); unit: Number of Adverse Events
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 27 | 14
Number of Adverse Events | 7.67 (8.23) | 5.29 (7.02)

8. Secondary Outcome: Headache Impact Test (HIT-6)
Description: Total Headache Impact Test (HIT-6) scores Pre-Treatment at Visit 2 vs. Post-Treatment (following final treatment), and at 1-Month Post-Treatment (Group A vs. Group B). HIT-6 is a series of 6 likert scale questions ranging from 1 to 5 with 1 being never and 5 being always. The HIT-6 answer options are weighted as follows: Never (1) = 6 points each, Rarely (2) = 9 points each, Sometimes (3) = 10 points each, Very often (4) = 11 points each, Always (5) = 13 points each. The total score for the HIT-6 ranges from 36 (subject answers all 6 questions as "Never") to 78 subject answers all 6 questions as "Always"), with higher total scores indicating more impact than lower scores, i.e., headaches cause greater impact on the subject's life.
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
units on a scale
  Pre-Treatment | 64.36 (4.93) | 64 (3.92)
  Post-Treatment | 59.85 (8.33) | 62.5 (4.96)
  1-Month Post-Treatment | 59.23 (8.97) | 61.92 (5.45)

9. Secondary Outcome: Overall Satisfaction
Description: Satisfaction scores Visit 2 vs. following treatment (Treatment 12) and at 1-Month Post-Treatment (Group A vs. Group B). Satisfaction scores are a likert scale ranging from 1 to 5 with 1 being complete dissatisfaction and 5 being complete satisfaction.
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marcaine | Saline
Number analyzed (Participants) | 26 | 12
units on a scale
  Visit 2 | 3.52 (0.75) | 3.00 (0.89)
  Following treatment (Treatment 12) | 3.55 (1.00) | 2.50 (0.97)
  1-Month Post-Treatment | 3.57 (0.99) | 2.64 (1.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent until study exit. The length of study participation was 34 weeks.
Groups:
- Marcaine: Marcaine (Group A) will receive treatment with 0.3 mL of 0.5% Marcaine delivered bilaterally with the Tx360™ device to the mucosa associated with the Sphenopalatine Ganglion (SPG)
  Marcaine: Marcaine used as a topical local anesthetic to block the SPG by delivering Marcaine directly to the specific area of mucosa associated with the SPG.
- Saline: Saline (Group B) will receive saline placebo delivered bilaterally with the Tx360TM device to the mucosa associated with the SPG.
Arm/Group | Marcaine | Saline
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/14
Other Adverse Events (participants affected / at risk) | 9/27 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marcaine (N=27) | Saline (N=14)
Pulmonary Embolism Resulting in Death (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marcaine (N=27) | Saline (N=14)
Bad Taste (General disorders) | 7 (30) | 1 (3)
Cold (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2)
Lacrimation (Eye disorders) | 8 (58) | 1 (1)
Mouth Numbness (General disorders) | 6 (37) | 0 (0)
Nasal Irritation (General disorders) | 4 (7) | 3 (6)
Dizziness (General disorders) | 0 (0) | 2 (5)
Ear Ringing (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Light Headedness (General disorders) | 1 (1) | 2 (3)
Sore Throat (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No